CLINICAL TRIAL: NCT04774809
Title: A Randomized, Double-blind, Vehicle-Controlled, Phase II/Ⅲ Seamless Adaptive Clinical Trail to Evaluate the Efficacy and Safety of SHR0302 Ointment in Adult Patients With Vitiligo
Brief Title: Assess the Efficacy and Safety of SHR0302 Ointment in Adult Patients With Vitiligo
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: terminated by sponsor
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSJ10828
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR0302 Low Dose (Active Comparator): Drug: SHR0302 SHR0302 Ointment BID Low Dose
  Interventions: Drug: Low Dose SHR0302 Ointment BID
- SHR0302 High Dose (Active Comparator): Drug: SHR0302 SHR0302 Ointment BID High Dose
  Interventions: Drug: High Dose SHR0302 Ointment BID
- Placebo Comparator: Vehicle (Placebo Comparator): Drug: vehicle Vehicle BID Placebo
  Interventions: Other: Placebo Comparator: Vehicle

INTERVENTIONS:
Drug: Low Dose SHR0302 Ointment BID — Low Dose SHR0302 Ointment BID
  Arms: SHR0302 Low Dose
Drug: High Dose SHR0302 Ointment BID — High Dose SHR0302 Ointment BID
  Arms: SHR0302 High Dose
Other: Placebo Comparator: Vehicle — Placebo
  Arms: Placebo Comparator: Vehicle

SUMMARY:
The purpose of this study is to assess the efficacy and safety of SHR0302 ointment in adult patients with Vitiligo.

DETAILED DESCRIPTION:
This study is a phase II/Ⅲ seamless adaptive clinical trial to evaluate the efficacy and safety of SHR0302 ointment in adult patients with non-segmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily signed an informed consent form.
2. Ages at ≥18 and ≤ 65 years
3. Clinical diagnosis of non-segmental vitiligo.
4. All women and men who are likely to give birth must be willing to use at least one efficient method of contraception from the signing of the informed consent form to 1 month after the last dose of IP.
5. Subjects who agree to discontinue all vitiligo-related treatments and camouflage cosmetics with therapeutic effect between screening visit and the last follow-up visit.
6. Subjects who are willing and able to comply with the scheduled visits and treatment plan, laboratory testing and other study procedures.

Exclusion Criteria:

1. Subjects who were diagnosed with segmental vitiligo, mixed vitiligo or unclassified vitiligo.
2. Subjects with historical or current evidence of clinically significant disease or lab test abnormalities or with disease that require the administration of prohibited drugs in this study.
3. Subjects with a malignant tumor or a history of malignant tumor (except for fully treated or resected skin non-metastatic basal cell carcinoma or squamous cell carcinoma).
4. Pregnant or lactating female subjects;
5. Subjects who have previously received JAK inhibitors therapy, systemic or oral
6. Subjects who had used any biologics within12 weeks before the baseline or 5 half-lives (whichever is longer).
7. Subjects who participated in other interventional clinical studies within 4 weeks before the baseline visit, or who were still within 5 half-lives of the last dose of the intervention clinical study drug at baseline.
8. Subjects who received a live or live-attenuated vaccination within 8 weeks before the baseline visit.
9. Any other condition that causes the subject to be unfit for the study as per discretion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Phase 2 | 24 weeks
  Phase 2: Percentage of change in face and neck vitiligo area scoring index (F-VASI) compared with baseline at week 24.
Phase 3 | 24 weeks
  Phase 3: Percentage of subjects whose face and neck vitiligo area scoring index improved by at least 75% (F-VASI75) compared with the baseline at week 24.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Wuhan No.1 Hospital, Wuhan, Hubei
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Xijing Hospital, Air Force Medical University, Xi'an, Shaanxi
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - West China School of Medicine, Chengdu, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - Hangzhou Third Hospital, Hangzhou, Zhejiang
  - Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - The First Hospital of Jillin University, Changchun
  - Sun. Yai- Sen Memorial Hospital, Sun. Yai- Sen University, Guangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Jiangsu Province Hospital, Nanjing
  - Huashan Hospital Affiliated To Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No